CLINICAL TRIAL: NCT06570135
Title: Brain Activity During Sexual Behavior in Patients With Primary Premature Ejaculation a Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KY20242242
Record Dates: First submitted 2024-07-29; First posted 2024-08-26 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-07

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- premature ejaculation group (Experimental)
  Interventions: Diagnostic Test: Detecting Brain Activity with Functional Near Infrared Spectroscopy
- Non-premature ejaculation group (Experimental)
  Interventions: Diagnostic Test: Detecting Brain Activity with Functional Near Infrared Spectroscopy

INTERVENTIONS:
Diagnostic Test: Detecting Brain Activity with Functional Near Infrared Spectroscopy — Use a functional near-infrared spectroscopy to detect brain activity in the two groups of subjects during resting state and task state.

SUMMARY:
This is a controlled study of patients with and without primary premature ejaculation. It is based on near-infrared spectroscopy (NIRS) functional brain imaging to detect and compare changes in brain activity in resting and task states (Simulated Sex) between the two groups of patients.

ELIGIBILITY:
Inclusion Criteria (primary premature ejaculation subjects):

* patients' age varied from 18 to 45 years；
* patients met the 2014 International Society for Sexual Medicine (ISSM) definition criteria for PPE；
* patients had a stable, heterosexual relationship with a single sexually active female partner for at least 6 months and with at least two sexual intercourses a week and kept stable during the study period;
* Patients with premature ejaculation lasting longer than 6 months；
* patients were identified if their scores were higher than 9 on the Chinese version of Premature Ejaculation Diagnostic Tool (PEDT);
* patients had no history of any previous therapies for PE or had recently stopped the therapies for at least 3 months
* patients had fully informed consent, signed informed consent form

Inclusion Criteria (Non-premature ejaculation subjects):

* Men between the ages of 18-45 years were included according to an age difference of <3 years between each patient and the primary premature ejaculation group, and if more than one volunteer was eligible at the same time, the one with the closest age was selected；
* Patient does not meet the 2014 International Society for Sexual Medicine (ISSM) criteria for defining premature ejaculation；
* patients had a stable, heterosexual relationship with a single sexually active female partner for at least 6 months and with at least two sexual intercourses a week and kept stable during the study period;
* patients had fully informed consent, signed informed consent form；

Exclusion Criteria:

* patients were diagnosed with secondary PE, variable PE, and subjective PE;
* patients were using medications for endocrinological, metabolic, chronic systemic, or psychiatric diseases;
* patients were abusing alcohol or illegal drugs；
* patients were diagnosed with erectile dysfunction (ED) if their scores were <21 on the abridged five-item International Index of Erectile Function (IIEF-5)
* patients were diagnosed with sexual hormone abnormalities, hyperthyroidism, hypothyroidism, Peyronie's disease, prostatitis, urethritis, or urinary tract infection;
* patients with head injuries that prevent them from completing near-infrared light brain function imaging
* Patients with severe schizophrenia, anxiety, depression or other neurological symptoms or poor compliance

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Results of near-infrared brain functional imaging | 1 hours
  Data on changes in oxygenated hemoglobin concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Air Force Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No